CLINICAL TRIAL: NCT03063138
Title: Evaluation of Three-dimensional Measurements of Wounds Using a Newly Developed 3D Camera
Brief Title: Evaluation of 3D Imaging Ulcer Camera
Acronym: 3D-DFU
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Line Bisgaard Jørgensen, MD, PhD student, Odense University Hospital
Other Study IDs: OUH3D03
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus; Diabetic Foot Ulcer; Wound; Chronic Disease
Keywords: Diabetic foot ulcer; Measurement; Wound healing; Measurement device; Three-dimensional measurements
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Wounds and Injuries; Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the intra- and inter-rater variability of wound measurements using the 3D camera and to compare with standard measurement methods (2D image method and gel injection). Forty-eight patients with wounds of various sizes are measured by four clinicians. Each wound is measured twice with the 3D camera, once by 2D image method and once by gel injection into wound cavity by two clinicians.

DETAILED DESCRIPTION:
Diabetic foot ulcers constitute an increasing health problem in Denmark concurrent with an ageing population and an increase in diabetes prevalence. Diabetic foot ulcers belong to the most serious and costly complications. Several studies have found that the size and depth of the wound is one of the major etiologic factors for delayed healing. Wound measurement is important in monitoring the healing process of wound and in evaluating the effect of treatment. Three-dimensional methods for measuring wound size have made it possible to evaluate the process of wound healing with respect to all dimensions. The investigators have developed a 3D camera, which is able to measure wound size (2D area, 3D area, perimeter and volume) and to assess wound characteristics.

The aim of the study is to evaluate the intra- and inter-rater variability of wound measurements using the 3D camera and to compare with standard measurement methods (2D image method and gel injection). Forty-eight patients with wounds of various sizes are measured by four clinicians. Each wound is measured twice with the 3D camera, once by 2D image method and once by gel injection into wound cavity by two clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients with wounds
* 18 years or older

Exclusion Criteria:

* Superficial ulcer (less than 5x5 mm with no substantial loss of subcutaneous tissue)
* Non-compliance (dementia, mental disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wounds from University Centre for Wound Healing, Odense University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Wound 2D area | 1 day
  Measured by 3D camera and 2D image method
Wound 3D area | 1 day
  Measured by 3D camera
Wound perimeter | 1 day
  Measured by 3D camera
Wound volume | 1 day
  Measured by 3D camera

CONTACTS AND LOCATIONS:
Overall Officials: Knud Yderstræde, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- University Centre of Wound Healing, Odense University Hospital (OUH), Odense, Denmark

IPD SHARING:
Plan to Share IPD: No